CLINICAL TRIAL: NCT07307066
Title: Real-Time Algorithm-Driven Ventilation Feedback to Improve Lung-Protective Ventilation in Critically Ill Patients
Acronym: REALVENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Hepingli Hospital (Unknown); Beijing No.6 Hospital (Unknown); Jinzhou Medical University (Other); Henan Provincial People's Hospital (Other); Binzhou Second People's Hospital (Unknown); Chongqing General Hospital (Other); Qujing Central Hospital of Yunnan Province (Unknown); Shandong Provincial Hospital (Other Government); Capital Medical University Affiliated Beijing Anzhen Hospital, Nanchong Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K6526
Record Dates: First submitted 2025-12-02; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: ARDS (Acute Respiratory Distress Syndrome); VILI (Ventilator-induced Lung Injury); Respiratory Failure; Critical Illness
MeSH Terms: conditions — Acute Lung Injury; Ventilator-Induced Lung Injury; Respiratory Insufficiency; Critical Illness

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the intervention arm or control arm. Intervention group Patients in the intervention arm will receive real-time ventilator waveform monitoring through the respiratory dynamics monitoring and feedback RemoteVentilate ViewTM system. The system continuously collects high-frequency waveform data (flow, pressure, volume) directly from the ventilator interface and analyses the following metrics: Tidal volume (VT) indexed to predicted body weight, Driving pressure (ΔP), Plateau pressure (Pplat), and Mechanical power (MP). Patient-ventilator asynchrony (PVA) events will be also collected in the system, including double triggering, ineffective efforts, reverse triggering, and flow starvation, ect.
  Control group The control group will receive standard ICU care, including routine monitoring of ventilator parameters such as tidal volume, plateau pressure, and oxygenation status. No structured feedback or external ventilation reports will be provided. This reflect
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, treating clinicians and bedside staff will not be blinded to group allocation. The real-time feedback reports and alerts generated by the respiratory dynamics monitoring and feedback RVV systemTM are inherently visible to the ICU team and require bedside review and interpretation, precluding clinician blinding. However, the following personnel will remain blinded to group allocation throughout the study: ①Outcome assessors (data analysts reviewing ventilator-free days, inflammatory biomarkers detection, VAP, barotrauma, mortality); ②The core biostatistical team responsible for primary and secondary outcome analyses; ③Members of the independent Data Monitoring Committee (DMC) reviewing interim safety data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REal-time Algorithm-driven Ventilation feedback to improve lung-protective ventilation in critically (Experimental): Patients in the intervention arm will receive real-time ventilator waveform monitoring through the respiratory dynamics monitoring and feedback RemoteVentilate ViewTM system. The system continuously collects high-frequency waveform data (flow, pressure, volume) directly from the ventilator interface and analyses the following metrics: Tidal volume (VT) indexed to predicted body weight, Driving pressure (ΔP), Plateau pressure (Pplat), and Mechanical power (MP). Patient-ventilator asynchrony (PVA) events will be also collected in the system, including double triggering, ineffective efforts, reverse triggering, and flow starvation, ect
  Interventions: Device: REal-time Algorithm-driven Ventilation feedback to improve lung-protective ventilation in critically
- Standard ICU care (Active Comparator): The control group will receive standard ICU care, including routine monitoring of ventilator parameters such as tidal volume, plateau pressure, and oxygenation status. No structured feedback or external ventilation reports will be provided. This reflects the prevailing standard of care in Chinese ICUs and is thus an appropriate comparator for assessing the added value of a real-time respiratory feedback platform.
  Interventions: Other: Standard ICU care

INTERVENTIONS:
Device: REal-time Algorithm-driven Ventilation feedback to improve lung-protective ventilation in critically — Patients in the intervention arm will receive real-time ventilator waveform monitoring through the respiratory dynamics monitoring and feedback RemoteVentilate ViewTM system. The system continuously collects high-frequency waveform data (flow, pressure, volume) directly from the ventilator interface and analyses the following metrics: Tidal volume (VT) indexed to predicted body weight, Driving pressure (ΔP), Plateau pressure (Pplat), and Mechanical power (MP). Patient-ventilator asynchrony (PVA) events will be also collected in the system, including double triggering, ineffective efforts, reverse triggering, and flow starvation, ect..
  Arms: REal-time Algorithm-driven Ventilation feedback to improve lung-protective ventilation in critically
Other: Standard ICU care — The control group will receive standard ICU care, including routine monitoring of ventilator parameters such as tidal volume, plateau pressure, and oxygenation status. No structured feedback or external ventilation reports will be provided. This reflects the prevailing standard of care in Chinese ICUs and is thus an appropriate comparator for assessing the added value of a real-time respiratory feedback platform.
  Arms: Standard ICU care

SUMMARY:
The REALVENT trial is designed to evaluate whether a real-time, algorithm-driven ventilation feedback strategy can improve lung-protective ventilation (LPV) achievement rates in critically ill patients receiving invasive mechanical ventilation. This multicentre randomised controlled trial will compare real-time respiratory waveform monitoring with automated feedback against standard ICU care. The primary endpoint is the LPV achievement rate over the first 72 hours.

DETAILED DESCRIPTION:
Mechanical ventilation is essential in modern intensive care but may cause ventilator-induced lung injury (VILI) when delivered with excessive tidal volume, airway pressure, or mechanical power, or in the presence of unrecognised patient-ventilator asynchrony. Despite guideline recommendations to limit tidal volume, plateau pressure, and driving pressure, real-world adherence to lung-protective ventilation (LPV) remains suboptimal, and clinicians often rely on intermittent, manual review of ventilator settings and waveforms.

The REALVENT trial tests a cloud-based respiratory dynamics monitoring and feedback system that continuously acquires high-frequency ventilator waveforms (pressure, flow, volume) and automatically computes key LPV metrics, including tidal volume indexed to predicted body weight, driving pressure, plateau pressure, mechanical power, and patient-ventilator asynchrony events. For patients in the intervention arm, the platform provides three layers of feedback over the first 72 hours after randomisation: (1) real-time alerts when LPV thresholds are exceeded; (2) 4-hour window indicator checks to capture sustained deviations; and (3) standardised 24-hour summary reports with recommendations for ventilator adjustment. These reports are reviewed by bedside clinicians and a central monitoring team, but all treatment decisions remain at the discretion of the local ICU team.

The control group receives usual care with standard bedside ventilator monitoring but without structured feedback from the platform. All other aspects of care, including fluid management, sedation, prone positioning, neuromuscular blockade, and adjunct respiratory monitoring (e.g., esophageal manometry or EIT), are left to clinician judgement and recorded.

The primary hypothesis is that algorithm-driven feedback will increase the proportion of time during the first 72 hours that all four LPV targets are simultaneously achieved compared with standard care. Secondary hypotheses are that improved LPV adherence will translate into more ventilator-free days, fewer ventilator-associated complications, lower inflammatory biomarker levels, and acceptable clinician workload and usability ratings.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Receiving invasive mechanical ventilation via endotracheal intubation at the time of screening
* Initiation of invasive mechanical ventilation within the past 24 hours
* PaO₂/FiO₂ ≤ 200 mmHg on PEEP ≥ 8 cmH₂O or, if arterial blood gas is unavailable: SpO₂/FiO₂ ≤ 235 with SpO₂ ≤ 97%
* Chest imaging (chest X-ray or CT) showing bilateral pulmonary infiltrates not fully explained by pleural effusions, lobar collapse, or pulmonary nodules
* Respiratory failure not fully explained by cardiac failure or fluid overload
* Expected to require invasive mechanical ventilation for ≥ 72 hours after enrollment

Exclusion Criteria:

* Receipt of extracorporeal membrane oxygenation (ECMO) or high-frequency oscillatory ventilation at screening
* Chronic ventilator dependence, defined as ≥ 21 consecutive days of mechanical ventilation prior to the current admission
* Brain death or anticipated withdrawal of life-sustaining treatment within 72 hours
* Pregnancy
* Known neuromuscular disease affecting spontaneous respiratory effort
* Prisoners or individuals unable to provide informed consent or surrogate consent
* Simultaneous enrollment in another interventional ICU study
* Lack of digital infrastructure for real-time ventilator waveform acquisition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The daily lung-protective ventilation achievement rate | Over the first 72 hours following randomisation
  The primary outcome is the daily lung-protective ventilation achievement rate over the first 72 hours following randomisation. Lung-protective ventilation is defined as simultaneous fulfilment of all of the following four criteria: Tidal volume (VT) < 8 mL/kg predicted body weight (PBW); Driving pressure (ΔP) < 15 cmH₂O; Plateau pressure (Pplat) < 30 cmH₂O; Mechanical power (MP) < 17 J/min. The daily achievement rate is calculated as the number of hours within each 24-hour period where all four targets are met, divided by 24, and expressed as a percentage. The mean of the three daily rates over the 72-hour period will be used as the primary outcome. This outcome reflects both physiological safety and clinician behaviour, and was selected based on its strong mechanistic link with ventilator-induced lung injury and previous observational data on variability in adherence

SECONDARY OUTCOMES:
Ventilator-free days at day 28 (VFD-28) | Day 28 after trial enrollment
  defined as the number of days alive and free from invasive mechanical ventilation between randomisation and day 28, with patients who die before day 28 considered as having 0 VFDs;
ICU length of stay | 28 days after ICU admission
  total number of days from ICU admission to ICU discharge;
Serum concentration of interleukin-1 beta (IL-1β) | Baseline (within 24hours) and 72 hours after trial enrollment
  Serum IL-1β concentration measured using standardized immunoassays.
Serum concentration of interleukin-6 (IL-6) | Baseline (within 24hours) and 72 hours after trial enrollment
  Serum IL-6 concentration measured using standardized immunoassays.
Serum concentration of soluble triggering receptor expressed on myeloid cells-1 (sTREM-1) | Baseline (within 24hours) and 72 hours after trial enrollment
  Serum sTREM-1 concentration measured using standardized immunoassays.
Incidence of ventilator-associated pneumonia (VAP) | 72 hours after trial enrollment
  based on CDC criteria, adjudicated by two independent reviewers;
Incidence of barotrauma | 72 hours after trial enrollment
  including pneumothorax, pneumomediastinum, or subcutaneous emphysema confirmed radiographically
ECMO initiation rate | 72 hours after trial enrollment
  proportion of patients who require extracorporeal support during the index ICU stay;
Mortality at day 28 | Day 28 after trial enrollment
  all-cause mortality;
Modified NASA Task Load Index (NASA-TLX) score (0-100) | 72 hours after trial enrollment
  Six-domain modified NASA-TLX; each domain rated 0-20; performance reverse-scored; mean transformed to 0-100; higher scores indicate greater perceived workload.
Clinician-reported usability score (mean of 5-item, 5-point Likert scale; range 1-5) | 72 hours after trial enrollment
  Five items rated 1-5; mean score reported; higher scores indicate better perceived usability.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the primary and secondary outcome results (including the final trial dataset and data dictionary) may be shared with qualified investigators for methodologically sound proposals, after publication of the main results and subject to institutional and ethical approvals. Data will be shared via secure data transfer agreements and will not contain any directly identifiable information.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available within one year of completion of the final follow up assessment, or within one year of primary manuscript publication, whichever comes first. Data will be available for 10 years.
Access Criteria: Outside investigators who wish to use data will submit a formal request, including rationale, analysis plan, and local Institutional Review Board (IRB) determination. Sponsor will review and respond to all requests. All data sharing will be codified by the appropriate contract / data use agreement. Recipient researchers must promise in writing to never attempt to access identifiable health/medical information or to attempt to identify the subject(s) who provided the specimen/data. Any intent to use materials or data for commercial purposes must be clearly disclosed as part of the request.

REFERENCES:
- [Result] Liu S, Zhao Z, Chen X, Chi Y, Yuan S, Cai F, Song Z, Ma Y, He H, Su L, Long Y. Evaluation of health care providers' ability to identify patient-ventilator triggering asynchrony in intensive care unit: a translational observational study in China. BMC Med Educ. 2025 Feb 4;25(1):182. doi: 10.1186/s12909-025-06638-5. PMID 39905371
- [Result] Chen X, Yuan S, Kassis EB, Zhang S, Chi Y, Liu S, Cai F, Ma Y, Li Y, Su L, Long Y. Methodological development of the remote ventilate view platform for real-time monitoring of patient-ventilator asynchrony and respiratory parameters in severe pneumonia patients. J Intensive Med. 2025 Sep 23;5(4):367-376. doi: 10.1016/j.jointm.2025.07.003. eCollection 2025 Oct. PMID 41180101
- [Result] Chen X, Fan J, Zhao W, Shi R, Guo N, Chang Z, Song M, Wang X, Chen Y, Li T, Li GG, Su L, Long Y; on bahalf of Beijing Dongcheng Critical Care Quality Control Centre Group. Application of a cloud platform that identifies patient-ventilator asynchrony and enables continuous monitoring of mechanical ventilation in intensive care unit. Heliyon. 2024 Jun 27;10(13):e33692. doi: 10.1016/j.heliyon.2024.e33692. eCollection 2024 Jul 15. PMID 39055813
- [Result] Su L, Lan Y, Chi Y, Cai F, Bai Z, Liu X, Huang X, Zhang S, Long Y. Establishment and Application of a Patient-Ventilator Asynchrony Remote Network Platform for ICU Mechanical Ventilation: A Retrospective Study. J Clin Med. 2023 Feb 16;12(4):1570. doi: 10.3390/jcm12041570. PMID 36836113